CLINICAL TRIAL: NCT02665221
Title: Single Center, Randomized, Open Label Study in Relapsing MS Patients on PLEGRIDY to Assess Topical Application of Preparation H (Phenylephrine) on Mitigation of Erythema Severity and Size.
Brief Title: Single Center, Open Label, Study of Preparation H on Erythema in Relapsing MS Patients Treated With PLEGRIDY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It was decided on 9/21/2016 to terminate this study early because LogPad devices the patients used to record their injection data was flawed
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-00173
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; erythema
MeSH Terms: conditions — Multiple Sclerosis; Erythema

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Other: No Treatment Arm
- Treatment group (Experimental)
  Interventions: Drug: Topical Preparation H arm

INTERVENTIONS:
Other: No Treatment Arm — Participants randomized to the control group will have no topical treatment at the injection site of the first full dose of Plegridy.
  Arms: Control group
Drug: Topical Preparation H arm — Preparation H (phenylephrine) treatment first full dose incidence injection site reaction.
  Arms: Treatment group

SUMMARY:
The primary purpose of this single center, randomized, open label study in relapsing Multiple Sclerosis (MS) patients on PLEGRIDY (peginterferon beta-1a) is to assess the effect of Preparation H (phenylephrine) Maximum Strength Cream compared to no topical treatment of injection site erythema after PLEGRIDY injection.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of relapsing multiple sclerosis, as defined by McDonald criteria.
* Age 18 to 70 years old, inclusive, at the time of informed consent.
* Naïve to PLEGRIDY or less than or equal to 12 months on PLEGRIDY therapy.

Exclusion Criteria:

* Primary progressive, secondary progressive or progressive relapsing MS.
* Concurrent enrollment in any clinical trial of an investigational product.
* Known allergy to any interferon or any component of PLEGRIDY (peginterferon beta-1a).
* Known allergy to phenylephrine, pramoxane or any component of Preparation H.
* History of hypersensitivity or intolerance to naproxen or acetaminophen (Tylenol) that would preclude the use of at least 1 of these during the study.
* History of inadequate response to subcutaneous interferon beta therapy.
* History of human immunodeficiency virus, hepatitis C virus antibody or current hepatitis B infection.
* History of premalignant and malignant disease including solid tumors and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured).
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
* History of seizure disorder or unexplained blackouts.
* History of suicidal ideation or an episode of clinically severe depression (as determined by the Investigator) within 3 months prior to Day 1.
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia), at the discretion of the Investigator, within 3 months prior to Day 1.
* History of drug or alcohol abuse (as defined by the Investigator) within 6 months prior to Day.
* Active bacterial or viral infection.
* Inability to comply with study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kalina, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 15 | 15
Completed | 0 | 0
Not Completed | 15 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 14 | 9 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Patient Erythema Self-Assessment (PSA) Score 6 hr After Application of Preparation H to First Injection Site Erythema Compared to Baseline PSA Score of Injection Site Erythema at Least 2 Hours After PLEGRIDY Injection.
Time Frame: 6 Hours
Population: Study was terminated. Logpad used by subjects was defective and data was not collected. No data analyzed.
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Width of Injection Site Erythema in Millimeters 6 hr After Application of Preparation H to First Injection Site Erythema Compared to Baseline Width of Injection Site Erythema at Least 2 Hours After Injection.
Description: Study was terminated. No data analyzed
Time Frame: 6 Hours
Population: Study was terminated. Logpad used by subjects was defective and data was not collected. No data analyzed.
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Patients Experiencing Injection Site Reaction Erythema, Itching and Pain.
Description: Study was terminated. No data analyzed. Study was terminated. No data analyzed because the Logpad being used by subjects was flawed.
Time Frame: 6 Hours
Population: Study was terminated. No data analyzed. Study was terminated. No data analyzed because the Logpad being used by subjects was flawed.
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Flu-like Symptom Scale at Last Visit Compared to Base Line.
Description: Study was terminated. No data analyzed because the Logpad being used by subjects was flawed.
Time Frame: 6 Hours
Population: Study was terminated. Logpad used by subjects was defective and data was not collected. No data analyzed.
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No